CLINICAL TRIAL: NCT03345732
Title: Intraoperative Evaluation Using Indocyanine Green and SPY Fluorescence Angiography to Prevent Wound Complications in Head and Neck Surgery Patients, an Observational Study
Brief Title: Intraoperative Evaluation Using ICG and SPY Fluorescence to Prevent Wound Complications in Head and Neck Surgery.
Status: Withdrawn | Type: Observational
Why Stopped: PI has been having difficulties obtaining ICG for this project.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-5976
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ICG and SPY system for wound complications

SUMMARY:
Wound complications, such as salivary-cutaneous fistulas and skin necrosis, result in significant patient morbidity and death. Head and neck wounds are complicated because of multiple tissue layers, critical structures and variable vascularity. When vascularity is compromised, wounds do not heal and can lead to life threatening haemorrhage or morbid infections. The field of microsurgical reconstruction has developed and expanded over the last 20 years to specifically ameliorate these issues. The challenge is that the vascularity of the microsurgical transplant or the recipient tissue bed can have areas of decreased vascularity that cannot be appreciated by the surgeon's intraoperative exam alone. Surgeons would be able to make better decisions with respect to the vascularity if there was an imaging technique that could indicate the vascular supply of the tissues undergoing surgical reconstruction.

Laser-assisted indocyanine green fluorescent dye angiography (LA-ICG) using the SPY System (Novadaq Technologies Inc., Richmond, British Columbia, Canada) is an intraoperative vascular imaging technique that improves the ability of a surgeon to assess the vascular supply in the surgical bed. This tool, which is approved by Health Canada for reconstructive surgery, has been used extensively in breast reconstruction and gastrointestinal procedures with encouraging results. The ability to address ischemic tissues intraoperatively could potentially decrease the rate of devastating wound complications in head and neck surgery patients. The objective of this observational study is to assess the effectiveness of LA-ICG in head and neck reconstructive procedures to reduce the rate of skin necrosis and fistula.

DETAILED DESCRIPTION:
This is a prospective, observational study in patients undergoing head and neck surgery with reconstruction. Patients will be identified preoperatively by the participating surgeons. Eligible patients will be >18 years of age with head and neck oncologic or traumatic reconstructive needs requiring surgical reconstruction of the soft tissues or bony structures of the head and neck who consent to use of ICG and the SPY System intraoperatively. Defect types to be included in the study are any hypopharyngeal defect (i.e. Total laryngectomy, total laryngectomy with partial pharyngectomy), tracheal defects, oral cavity defects at risk for devascularized mucosa, or large skin defects requiring rotation-advancement flaps for closure. Donor types to be included are pedicled locoregional muscle flaps including pectoralis muscle flaps, cervicofacial skin advancement flaps, infrascapular and suprascapular flaps, and any free flap used to reconstruct the defects mentioned previously.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years old) who are undergoing reconstruction for traumatic or oncologic head and neck wounds
2. Specific defects eligible are any pharyngeal, tracheal, or oral cavity defects at risk of devascularized mucosa, or large skin defects requiring skin advancement flaps. This includes laryngectomy/laryngectomy-partial pharyngectomy with primary closure.
3. Patient with the above defects that will be having reconstruction with the following donor tissues: local, regional or autogenous free flaps.
4. Informed consent

Exclusion Criteria:

1. Patients who are pregnant or nursing
2. Patients with an allergy to iodine (contrast ICG dye contains sodium iodide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer requiring surgery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12-08 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
ICG/SPY system for tissue viability | introperatively
  To determine how often ICG/SPY system can be used to determine debridement of recipient or donor tissue during head and neck reconstruction

SECONDARY OUTCOMES:
Amount of tissue debridement | intraoperatively
  To determine how much tissue is debrided; and how often flap design is altered due to findings of the SPY system

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada